CLINICAL TRIAL: NCT00757159
Title: Randomised, Clinical Controlled Study on Treatment of Intra-bony Defects With Enamel Matrix Protein (Emdogain®) vs. Nanocrystalline Hydroxyapatite (Ostim®)
Brief Title: Study on Regenerative Treatment of Intra-bony Defects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZER-PA_01-2008
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Periodontal Disease; Periodontal Attachment Loss
Keywords: Periodontal disease; Hydroxyapatite; Enamel matrix protein; Regeneration; Human
MeSH Terms: conditions — Periodontal Diseases; Periodontal Attachment Loss

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Device: Ostim
- 2 (Active Comparator)
  Interventions: Device: Emdogain

INTERVENTIONS:
Device: Ostim — Ostim® is synthetically manufactured and comprises nanocrystalline hydroxyapatite. The small particle size facilitates resorption. Ostim is an aqueous watery paste and can be used to fill bone defects or to build up bony structures in the region of the jaws. Ostim is osteoconductive, facilitating bone growth. It will act as a scaffolding for the new bone. Ostim is absorbed during the healing process, in the beginning it is osseously interweaved and finally replaced by natural bone.
  Other Names: synthetic hydroxyapatite
  Arms: 1
Device: Emdogain — Emdogain® consists of sterile lyophilised Enamel Matrix Derivative with sterile aqueous solution of Propylene Glycol Alginate, 30 mg/ml.
  Other Names: enamel matrix protein
  Arms: 2

SUMMARY:
The aim of this investigation is to determine whether a synthetic hydroxyapatite is as effective as an enamel matrix protein for periodontal regeneration in patients who have intra-bony periodontal defects.

DETAILED DESCRIPTION:
Regeneration of periodontal tissues that have been diminished by periodontal disease is the main goal of periodontal therapy. While conventional surgical therapy only offers limited potential towards recovering tooth-supporting tissues, more recently developed techniques lead to a greater and more predictable regeneration of the periodontal structures. Among these techniques, application of enamel matrix proteins or bone grafts can promote periodontal regeneration.

The study is a prospective, controlled, mono-center, randomized, clinical trial, that is open to the operator, blinded to the examiner. It will be conducted in a parallel group design. Participants who have at least 1 intra-bony periodontal defect will receive regenerative surgery at baseline with the randomly selected devices. A newly developed synthetically manufactured bone grafting material made of hydroxyapatite (Ostim) will be the product under investigation. An enamel matrix protein derivative (Emdogain) will act as control device. Both materials will be applied in intra-bony defects during periodontal flap surgery. Follow-ups will take place at 7 and 14 days post surgery, and at 3, 6, 9, and 12 months.

The primary aim is to compare the effectiveness of the test product with the control in the treatment of 1- and 2-wall intrabony periodontal defects on the amount of bone fill 12 months after surgery. Secondary parameters will be the clinical attachment level gain and reduction of probing pocket depth at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged between 18 and 70 years.
* Presence of at least one 1- or 2-wall intrabony periodontal defect.
* Defect width at least 2 mm.
* Defect depth at least 4 mm.
* Defect located at a single rooted tooth or at the approximal site of a multi-rooted tooth if the tooth is not affected by a furcation involvement.
* Written informed consent.
* Subject must be judged healthy by the investigator at the time of surgery.
* Subjects must have had a plaque index < 0.8 at the end of the initial periodontal therapy.

Exclusion Criteria:

* Medical conditions required prolonged use of steroids.
* Standard blood tests performed by the medical practitioner showing leukocyte dysfunction and deficiencies.
* History of haemophilia, bleeding disorders, or cumarin therapy.
* History of neoplastic disease requiring the use of chemotherapy.
* History of radiation therapy of the head and neck.
* History of renal failure or chronic renal diseases.
* Chronic liver diseases.
* Severe or uncontrolled metabolic bone disorders.
* Uncontrolled endocrine disorders (including diabetes).
* Current pregnancy at the time of recruitment.
* Physical handicaps that would interfere with the ability to perform adequate oral hygiene.
* Use of any investigational drug or device within the 90 day period prior to surgery on study day 0.
* Alcoholism or chronical drug abuse.
* Immuno-compromised patients (including HIV).
* Smokers (occasional smoking is allowed).
* Conditions or circumstances , in the opinion of the investigator, that could represent a general contra-indication for surgical procedures or would prevent completion of study participation or interfere with analysis of study results, such as a history of non-compliance, or unreliability.
* Local inflammation.
* Mucosal diseases (e.g. erosive lichen planus).
* History of local radiation therapy.
* Presence of oral lesions (e.g. ulceration, malignancy).
* Inadequate oral hygiene or patient who is unmotivated for home care.
* Teeth with untreated endodontic or cariologic problems.
* Defects that during surgery show deviation from the inclusion criteria.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Amount of bone fill after surgery | 12 months

SECONDARY OUTCOMES:
Clinical attachment level gain and reduction of probing pocket depth | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hoffmann, Prof., Principal Investigator — Technische Universität Dresden
Locations (1):
- Dresden University of Technology, Dental School, Department of Conservative Dentistry, Dresden, Germany

REFERENCES:
- [Derived] Al Machot E, Hoffmann T, Lorenz K, Khalili I, Noack B. Clinical outcomes after treatment of periodontal intrabony defects with nanocrystalline hydroxyapatite (Ostim) or enamel matrix derivatives (Emdogain): a randomized controlled clinical trial. Biomed Res Int. 2014;2014:786353. doi: 10.1155/2014/786353. Epub 2014 Feb 9. PMID 24689056